CLINICAL TRIAL: NCT02255409
Title: A Phase III, Randomized, Observer Blind, Multicenter Study to Evaluate the Safety and Immunogenicity of Repeated Exposure to an Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV), Administered to Subjects Previously Vaccinated in Trial V118_05
Brief Title: Clinical Study to Evaluate Safety, Immunogenicity of Investigational Flu Vaccine Compared to an Approved Flu Vaccine (QIV) in Children Previously Vaccinated in Trial V118_05
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V118_05E1; 2014-002599-95 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- aQIV (Experimental): Adjuvanted Quadrivalent Subunit Influenza
  Interventions: Biological: Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV)
- QIV (Active Comparator): Non-Adjuvanted Quadrivalent Subunit Influenza
  Interventions: Biological: non-adjuvanted Quadrivalent Influenza Vaccine (QIV)

INTERVENTIONS:
Biological: Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV) — 1 dose 0.25 ml: ≥6 months to <36 months, 0.5 ml: ≥36 months to <72 months
  Arms: aQIV
Biological: non-adjuvanted Quadrivalent Influenza Vaccine (QIV) — 1 dose 0.25 ml: ≥6 months to <36 months, 0.5 ml: ≥36 months to <72 months
  Arms: QIV

SUMMARY:
Safety, Immunogenicity of an Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine Compared to Non-Adjuvanted Comparator Influenza Vaccine in Children Previously Vaccinated in Trial V118_05

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject who has completed their Day 181 clinic visit for non-naïve subjects or their Day 209 clinic visit for naïve subjects in parent study.
2. Individuals who give written informed consent, who can comply with study procedures, and who are available for follow-up

Exclusion Criteria:

1. Individuals recently vaccinated against influenza.
2. Subjects with contraindications to receive influenza vaccine.
3. Please contact the site for additional eligibility criteria.

Ages: 12 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 607 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (17):
  - San Diego, California
  - San Gabriel, California
  - Colorado Springs, Colorado
  - Melbourne, Florida
  - Augusta, Kansas
  - Newton, Kansas
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Bellevue, Nebraska
  - Binghamton, New York
  - Dayton, Ohio
  - Austin, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
- Finland (8):
  - Espoo
  - Helsinki
  - Jarvenpaa
  - Kokkola
  - Pori
  - Tampere
  - Turku
  - Vantaa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 30 sites in 2 countries (Finland and United States)
Pre-assignment Details: All enrolled subjects were included in the trial
Groups:
- Adjuvanted Quadrivalent Influenza Vaccine (aQIV): Subjects approximately ≥12 months to 7 years of age who had received aQIV in the parent study V118_05 received aQIV in study V118_05E1.
- Comparator Quadrivalent Influenza Vaccine (QIV): Subjects approximately ≥12 months to 7 years of age who had received TIV in the parent study V118_05 received QIV in study V118_05E1.
Period: Overall Study
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Started | 318 | 289
Completed | 304 | 258
Not Completed | 14 | 31
Not completed — Administrative Reason | 3 | 7
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 10 | 19

BASELINE CHARACTERISTICS:
Groups:
- Adjuvanted Quadrivalent Influenza Vaccine (aQIV): Subjects approximately ≥12 months to 7 years of age who had received aQIV in the parent study V118_05 received aQIV in the study V118_05E1.
- Total: Total of all reporting groups
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV) | Total
Number analyzed (Participants) | 318 | 289 | 607
Age, Continuous [Mean (Standard Deviation); unit: months] | 44.7 (19.04) | 42.0 (17.47) | 43.4 (18.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 155 | 326
  Male | 147 | 134 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 48 | 112
  Not Hispanic or Latino | 253 | 241 | 494
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 75 | 65 | 140
  White | 231 | 209 | 440
  More than one race | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 269 | 238 | 507
  Finland | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Number of Subjects With SAEs, AEs Leading to Withdrawal From the Study, NOCDs, AESIs and Medically Attended AEs.
Description: Safety was assessed in terms of number of subjects between 12 months and 7 years of age reporting unsolicited events up to 12 months after last vaccination with either aQIV or QIV (comparator): serious adverse events (SAEs), AEs leading to study withdrawal, new onset chronic disease (NOCDs), adverse events of special interest (AESIs) and medically attended AEs after vaccination.
Time Frame: Day 1 through Day 356
Population: The Unsolicited Safety Set consisting of subjects who received a study vaccination and who had any AE assessments (ie, a subject did not have to have an AE to be included in this population) was used for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- aQIV: Subjects approximately ≥12 months to 7 years of age who had received aQIV in the parent study V118_05 received aQIV in study V118_05E1.
- Comparator QIV: Subjects approximately ≥12 months to 7 years of age who had received TIV in the parent study V118_05 received QIV in study V118_05E1.
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 317 | 288
Participants
  SAEs | 7 | 4
  At least possibly related SAEs | 0 | 0
  NOCDs | 13 | 7
  AESIs | 1 | 1
  Medically attended AEs | 161 | 141
  AEs leading to withdrawal | 0 | 0

2. Primary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion and Differences in Percentage of Subjects Achieving Seroconversion for Homologous Influenza Strains (Day 22)
Description: The percentage of subjects achieving seroconversion at Day 22 after vaccination is reported for homologous strains; Seroconversion is defined as hemagglutination inhibition (HI) ≥1:40 for subjects negative at baseline [<1:10]; or a minimum 4-fold increase in HI titer for subjects positive at baseline [HI ≥1:10]; Strains tested: A/H1N1 is Influenza A H1N1 California/7/2009 Egg Ab; A/H3N2 is Influenza A H3N2 Texas/50/2012 Ab; B/Yamagata is Influenza B Massachusetts/2/2012 Ab; B/Victoria is Influenza B Brisbane/60/2008 Egg Ab
Time Frame: Day 1, Day 22
Population: The Full Analysis Set for Immunogenicity consisting of all enrolled subjects who received a study vaccination and provided evaluable serum samples (homologous strains) for both before (baseline) and after vaccination (ie, Day 22 and/or Day 181).
  Day 22 analyses are reported for the 302 and 257 (256 for the A/H3N2 strain) participants in the aQIV and Comparator QIV groups, respectively, who had immunogenicity data at both Day 1 and Day 22.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 302 | 257
Percentage of subjects
  A/H1N1 | 57.9 [52.2 to 63.6] | 56.4 [50.1 to 62.6]
  A/H3N2: number analyzed (Participants) | 302 | 256
  A/H3N2 | 50.7 [44.9 to 56.4] | 56.6 [50.3 to 62.8]
  B/Yamagata | 73.5 [68.2 to 78.4] | 57.2 [50.9 to 63.3]
  B/Victoria | 72.2 [66.8 to 77.2] | 58.0 [51.7 to 64.1]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; Vaccine Group Difference (aQIV - QIV) for A/H1N1 at Day 22; Test type: Other; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-6.7 to 9.7]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; Vaccine Group Difference (aQIV - QIV) for A/H3N2 at Day 22; Test type: Other; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-14.2 to 2.3]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; Vaccine Group Difference (aQIV - QIV) for B/Yamagata at Day 22; Test type: Other; Mean Difference (Final Values) = 16.3, 95% CI 2-sided [8.4 to 24.1]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; Vaccine Group Difference (aQIV - QIV) for B/Victoria at Day 22; Test type: Other; Mean Difference (Final Values) = 14.2, 95% CI 2-sided [6.3 to 22.0]

3. Primary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving HI Titer ≥ 1:40 and and Differences in Percentage of Subjects Achieving HI Titer ≥ 1:40 for Homologous Influenza Strains (Day 22).
Description: The percentage of subjects achieving HI titer ≥1:40 at Day 22 after vaccination is reported for homologous strains. Strains tested: A/H1N1 is Influenza A H1N1 California/7/2009 Egg Ab; A/H3N2 is Influenza A H3N2 Texas/50/2012 Ab; B/Yamagata is Influenza B Massachusetts/2/2012 Ab; B/Victoria is Influenza B Brisbane/60/2008 Egg Ab
Time Frame: Day 1, Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Comparator Quadrivalent Influenza Vaccine (QIV): Subjects approximately ≥12 months to 7 years of age who had received TIV in the parent study V118_05 received QIV in the study V118_05E1.
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 302 | 257
Percentage of subjects
  A/H1N1, Homologous | 100.0 [98.8 to 100.0] | 99.6 [97.9 to 100.0]
  A/H3N2, Homologous: number analyzed (Participants) | 302 | 256
  A/H3N2, Homologous | 99.7 [98.2 to 100.0] | 100.0 [98.6 to 100.0]
  B/Yamagata, Homologous | 95.7 [92.8 to 97.7] | 81.3 [76.0 to 85.9]
  B/Victoria, Homologous | 98.0 [95.7 to 99.3] | 72.0 [66.1 to 77.4]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H1N1 at Day 22; Test type: Other; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.9 to 2.2]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H3N2 at Day 22; Test type: Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.9 to 1.2]
Statistical Analysis 3: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Yamagata at Day 22; Test type: Other; Mean Difference (Final Values) = 14.4, 95% CI 2-sided [9.3 to 20.0]
Statistical Analysis 4: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Victoria at Day 22; Test type: Other; Mean Difference (Final Values) = 26.0, 95% CI 2-sided [20.6 to 32.0]

4. Secondary Outcome: Safety Endpoint: Number of Subjects With a Diagnosis of Failure to Thrive or Short Stature
Description: Short stature was defined as a height/length that was 2 or more standard deviations below the mean for age and gender within a population and was assessed as being below the 2nd z-score (worse outcome) on the length/height-for-age scale. Failure-to-thrive was defined by inadequate weight gain and physical growth and assessed through 2 or more of the following criteria: height/length-for-age, weight-for-age or weight-for-height/length below the 2nd z-score, a child's growth line crossing a z-score line, a sharp change in growth curve or a curve that remains flat. The observations were made for 2 or more time points each divided by at least 2 months.
Time Frame: Day 1 through Day 366 (Day 1, Day 22, Day 181, Day 366)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 317 | 290
participants
  Subjects with diagnosis of failure to thrive | 0 | 0
  Subjects with diagnosis of short stature | 0 | 0

5. Secondary Outcome: Safety Endpoint: Number of Subjects With Any Unsolicited AEs
Description: Safety was assessed in terms of number of subjects between 12 months and 7 years of age reporting unsolicited events up to 12 months after last vaccination with either aQIV or QIV (comparator).
Time Frame: Day 1 through Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Comparator QIV: Subjects approximately ≥12 months to 7 years of age who had received TIV in the parent study V118_05 received QIV in the present study V118_05E1.
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 317 | 288
Participants | 85 | 60

6. Secondary Outcome: Safety Endpoint: Number of Subjects With Solicited Local and Systemic Adverse Events (AEs)
Description: Safety was assessed in terms of number of subjects between 12 months and 7 years of age reporting solicited local and systemic AEs, day 1 to day 7 after vaccination with either aQIV or QIV (comparator).
Time Frame: Up to 7 days following vaccination
Population: The Solicited Safety Set consisting of subjects who received a study vaccination and had any assessment of local and systemic reactions and/or assessment of any use of analgesics/antipyretics was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 317 | 288
Participants
  Solicited AEs, Any | 202 | 148
  Solicited Local AEs | 173 | 112
  Solicited Systemic AEs | 127 | 80
  Other | 66 | 26

7. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion and Differences in Percentage of Subjects Achieving Seroconversion for Homologous Influenza Strains (Day 181)
Description: The percentage of subjects achieving seroconversion at Day 181 after vaccination is reported for homologous strains. Seroconversion is defined as HI ≥1:40 for subjects negative at baseline [<1:10]; or a minimum 4-fold increase in HI titer for subjects positive at baseline [HI ≥1:10]; Strains tested: A/H1N1 is Influenza A H1N1 California/7/2009 Egg Ab; A/H3N2 is Influenza A H3N2 Texas/50/2012 Ab; B/Yamagata is Influenza B Massachusetts/2/2012 Ab; B/Victoria is Influenza B Brisbane/60/2008 Egg Ab.
Time Frame: Day 1, Day 181
Population: The Full Analysis Set for Immunogenicity consisting of all enrolled subjects who received a study vaccination and provided evaluable serum samples (homologous strains) for both before (baseline) and after vaccination (ie, Day 22 and/or Day 181).
  Day 181 analyses are reported for the 289 and 251 participants in the aQIV and Comparator QIV groups, respectively, who had immunogenicity data at both Day 1 and Day 181.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 289 | 251
Percentage of subjects
  A/H1N1, Homologous | 27.7 [22.6 to 33.2] | 21.9 [17.0 to 27.5]
  A/H3N2, Homologous | 30.1 [24.9 to 35.8] | 27.9 [22.4 to 33.9]
  B/Yamagata, Homologous | 24.6 [19.7 to 29.9] | 12.7 [8.9 to 17.5]
  B/Victoria, Homologous | 21.5 [16.9 to 26.6] | 22.7 [17.7 to 28.4]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H1N1 at Day 181; Test type: Other; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-1.6 to 13.0]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H3N2 at Day 181; Test type: Other; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-5.5 to 9.8]
Statistical Analysis 3: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Yamagata at Day 181; Test type: Other; Mean Difference (Final Values) = 11.8, 95% CI 2-sided [5.3 to 18.3]
Statistical Analysis 4: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Victoria at Day 181; Test type: Other; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-8.4 to 5.7]

8. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving HI Titer ≥ 1:40 and Difference in Percentage of Subjects Achieving HI Titer ≥ 1:40 for Homologous Influenza Strains (Day 181)
Description: The percentage of subjects achieving HI titer ≥1:40 at Day 181 after vaccination is reported for homologous strains; Strains tested: A/H1N1 is Influenza A H1N1 California/7/2009 Egg Ab; A/H3N2 is Influenza A H3N2 Texas/50/2012 Ab; B/Yamagata is Influenza B Massachusetts/2/2012 Ab; B/Victoria is Influenza B Brisbane/60/2008 Egg Ab
Time Frame: Day 1, Day 181
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 289 | 251
Percentage of subjects
  A/H1N1, Homologous | 99.7 [98.1 to 100.0] | 94.8 [91.3 to 97.2]
  A/H3N2, Homologous | 99.7 [98.1 to 100.0] | 94.0 [90.3 to 96.6]
  B/Yamagata, Homologous | 73.0 [67.5 to 78.0] | 39.8 [33.7 to 46.2]
  B/Victoria, Homologous | 82.4 [77.5 to 86.6] | 45.0 [38.8 to 51.4]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H1N1 at Day 181; Test type: Other; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [2.4 to 8.4]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H3N2 at Day 181; Test type: Other; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [3.1 to 9.3]
Statistical Analysis 3: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Yamagata at Day 181; Test type: Other; Mean Difference (Final Values) = 33.2, 95% CI 2-sided [25.0 to 40.9]
Statistical Analysis 4: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Victoria at Day 181; Test type: Other; Mean Difference (Final Values) = 37.3, 95% CI 2-sided [29.6 to 44.7]

9. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean HI Titers (GMTs) and GMT Ratios for Homologous Influenza Strains (Day 1, Day 22, Day 181)
Description: Adjusted GMT, GMR and 95% confidence interval (CI) were analyzed using ANCOVA with study specific covariates. Strains tested: A/H1N1 is Influenza A H1N1 California/7/2009 Egg Ab; A/H3N2 is Influenza A H3N2 Texas/50/2012 Ab; B/Yamagata is Influenza B Massachusetts/2/2012 Ab; B/Victoria is Influenza B Brisbane/60/2008 Egg Ab
Time Frame: Day 1, Day 22, Day 181
Population: The Full Analysis Set for Immunogenicity consisting of all enrolled subjects who received a study vaccination and provided evaluable serum samples (homologous strains) for both before (baseline) and after vaccination (ie, Day 22 and/or Day 181).
  Day 22 analyses are reported for 302 and 257 (256 for the A/H3N2 strain) participants in the aQIV and Comparator QIV groups, respectively.
  Day 181 analyses are reported for 289 and 251 participants in the aQIV and Comparator QIV groups, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 309 | 273
titer
  Day 1: A/H1N1, Homologous | 320.27 [261.9 to 391.6] | 165.23 [134.0 to 203.8]
  Day 22: A/H1N1, Homologous: number analyzed (Participants) | 302 | 257
  Day 22: A/H1N1, Homologous | 1036.27 [923.2 to 1163.2] | 700.78 [623.7 to 787.3]
  Day 181: A/H1N1, Homologous: number analyzed (Participants) | 289 | 251
  Day 181: A/H1N1, Homologous | 424.00 [374.2 to 480.5] | 282.31 [248.8 to 320.4]
  Day 1: A/H3N2, Homologous | 336.88 [268.5 to 422.7] | 155.97 [123.1 to 197.6]
  Day 22: A/H3N2, Homologous: number analyzed (Participants) | 302 | 256
  Day 22: A/H3N2, Homologous | 1221.47 [1093.1 to 1364.9] | 908.63 [810.0 to 1019.3]
  Day 181: A/H3N2, Homologous: number analyzed (Participants) | 289 | 251
  Day 181: A/H3N2, Homologous | 611.09 [529.0 to 705.9] | 454.46 [391.5 to 527.6]
  Day 1: B/Yamagata, Homologous | 32.36 [26.9 to 38.9] | 17.78 [14.7 to 21.5]
  Day 22: B/Yamagata, Homologous: number analyzed (Participants) | 302 | 257
  Day 22: B/Yamagata, Homologous | 176.04 [150.8 to 205.5] | 100.80 [86.1 to 181.1]
  Day 181: B/Yamagata, Homologous: number analyzed (Participants) | 289 | 251
  Day 181: B/Yamagata, Homologous | 54.08 [46.6 to 62.8] | 29.26 [25.1 to 34.1]
  Day 1: B/Victoria, Homologous | 46.41 [38.0 to 56.6] | 14.33 [11.6 to 17.6]
  Day 22: B/Victoria, Homologous: number analyzed (Participants) | 302 | 257
  Day 22: B/Victoria, Homologous | 244.52 [203.6 to 293.7] | 163.95 [135.6 to 198.2]
  Day 181: B/Victoria, Homologous: number analyzed (Participants) | 289 | 251
  Day 181: B/Victoria, Homologous | 65.85 [55.9 to 77.6] | 50.88 [42.9 to 60.3]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); The ratio of GMT (GMTr) values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H1N1 at Day 1; Test type: Other; GMT Ratio = 1.94, 95% CI 2-sided [1.6 to 2.4]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H1N1 at Day 22; Test type: Other; GMT Ratio = 1.48, 95% CI 2-sided [1.3 to 1.7]
Statistical Analysis 3: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H1N1 at Day 181; Test type: Other; GMT Ratio = 1.50, 95% CI 2-sided [1.3 to 1.7]
Statistical Analysis 4: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 1; Test type: Other; GMT Ratio = 2.16, 95% CI 2-sided [1.7 to 2.7]
Statistical Analysis 5: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 22; Test type: Other; GMT Ratio = 1.34, 95% CI 2-sided [1.2 to 1.5]
Statistical Analysis 6: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 181; Test type: Other; GMT Ratio = 1.34, 95% CI 2-sided [1.2 to 1.6]
Statistical Analysis 7: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Yamagata at Day 1; Test type: Other; GMT Ratio = 1.82, 95% CI 2-sided [1.5 to 2.2]
Statistical Analysis 8: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Yamagata at Day 22; Test type: Other; GMT Ratio = 1.75, 95% CI 2-sided [1.5 to 2.0]
Statistical Analysis 9: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Yamagata at Day 181; Test type: Other; GMT Ratio = 1.85, 95% CI 2-sided [1.6 to 2.2]
Statistical Analysis 10: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Victoria at Day 1; Test type: Other; GMT Ratio = 3.24, 95% CI 2-sided [2.7 to 4.0]
Statistical Analysis 11: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Victoria at Day 22; Test type: Other; GMT Ratio = 1.49, 95% CI 2-sided [1.2 to 1.8]
Statistical Analysis 12: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Victoria at Day 181; Test type: Other; GMT Ratio = 1.29, 95% CI 2-sided [1.1 to 1.5]

10. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratios (GMR) for Homologous Influenza Strains
Description: The GMR is the geometric mean of the fold increase in HI titer from Day 1 to Day 22 or Day 181. Adjusted GMT, GMR and 95% CI were analyzed using ANCOVA with study specific covariates. Strains tested: A/H1N1 is Influenza A H1N1 California/7/2009 Egg Ab; A/H3N2 is Influenza A H3N2 Texas/50/2012 Ab; B/Yamagata is Influenza B Massachusetts/2/2012 Ab; B/Victoria is Influenza B Brisbane/60/2008 Egg Ab
Time Frame: Day 1, Day 22, and Day 181
Population: The Full Analysis Set for Immunogenicity consisting of all enrolled subjects who received a study vaccination and provided evaluable serum samples (homologous strains) for both before (baseline) and after vaccination (ie, Day 22 and/or Day 181).
  Note: Subjects may be included in the Day 181 analyses but not the Day 22 analyses (and vice versa).
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 309 | 273
ratio
  Day 22/Day 1: A/H1N1, Homologous: number analyzed (Participants) | 302 | 257
  Day 22/Day 1: A/H1N1, Homologous | 5.82 [5.2 to 6.5] | 3.93 [3.5 to 4.4]
  Day 181/Day 1: A/H1N1, Homologous: number analyzed (Participants) | 289 | 251
  Day 181/Day 1: A/H1N1, Homologous | 2.40 [2.1 to 2.7] | 1.60 [1.4 to 1.8]
  Day 22/Day 1: A/H3N2, Homologous: number analyzed (Participants) | 302 | 257
  Day 22/Day 1: A/H3N2, Homologous | 5.41 [4.8 to 6.0] | 4.03 [3.6 to 4.5]
  Day 181/Day 1: A/H3N2, Homologous: number analyzed (Participants) | 289 | 251
  Day 181/Day 1: A/H3N2, Homologous | 2.73 [2.4 to 3.2] | 2.03 [1.8 to 2.4]
  Day 22/Day 1: B/Yamagata, Homologous: number analyzed (Participants) | 302 | 257
  Day 22/Day 1: B/Yamagata, Homologous | 8.33 [7.1 to 9.7] | 4.77 [4.1 to 5.6]
  Day 181/Day 1: B/Yamagata, Homologous: number analyzed (Participants) | 289 | 251
  Day 181/Day 1: B/Yamagata, Homologous | 2.57 [2.2 to 3.0] | 1.39 [1.2 to 1.6]
  Day 22/Day 1: B/Victoria, Homologous: number analyzed (Participants) | 302 | 257
  Day 22/Day 1: B/Victoria, Homologous | 9.26 [7.7 to 11.1] | 6.21 [5.1 to 7.5]
  Day 181/Day 1: B/Victoria, Homologous: number analyzed (Participants) | 289 | 251
  Day 181/Day 1: B/Victoria, Homologous | 2.55 [2.2 to 3.0] | 1.97 [1.7 to 2.3]

11. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion and Difference in Percentage of Subjects Achieving Seroconversion for Heterologous Influenza Strains (Day 181)
Description: The percentage of subjects achieving seroconversion at Day 181 after vaccination is reported for homologous strains. Seroconversion is defined as HI ≥1:40 for subjects negative at baseline [<1:10]; or a minimum 4-fold increase in HI titer for subjects positive at baseline [HI ≥1:10]; Strains tested: A/H3N2 is Influenza A H3N2 Hong Kong/2014 Ab; B/Yamagata is Influenza B Phuket/2013 Ab
Time Frame: Day 1, Day 181
Population: The Full Analysis Set for Immunogenicity consisting of all enrolled subjects who received a study vaccination and provided evaluable serum samples (heterologous strains) for both before (baseline) and after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 155 | 138
Percentage of subjects
  A/H3N2, Heterologous | 36.1 [28.6 to 44.2] | 30.4 [22.9 to 38.8]
  B/Yamagata, Heterologous: number analyzed (Participants) | 155 | 136
  B/Yamagata, Heterologous | 27.7 [20.9 to 35.5] | 13.2 [8.0 to 20.1]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H3N2 at Day 181; Test type: Other; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-5.2 to 16.3]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Yamagata at Day 181; Test type: Other; Mean Difference (Final Values) = 14.5, 95% CI 2-sided [5.3 to 23.6]

12. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving HI Titer ≥ 1:40 and Difference in Percentage of Subjects Achieving HI Titer ≥ 1:40 for Heterologous Influenza Strains (Day 181)
Description: The percentage of subjects achieving HI titer ≥1:40 at Day 181 after vaccination is reported for homologous strains; Strains tested: A/H3N2 is Influenza A H3N2 Hong Kong/2014 Ab; B/Yamagata is Influenza B Phuket/2013 Ab
Time Frame: Day 1, Day 181
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 155 | 138
Percentage of subjects
  A/H3N2, Heterologous | 96.8 [92.6 to 98.9] | 80.4 [72.8 to 86.7]
  B/Yamagata, Heterologous: number analyzed (Participants) | 155 | 136
  B/Yamagata, Heterologous | 83.9 [77.1 to 89.3] | 37.5 [29.4 to 46.2]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for A/H3N2 at Day 181; Test type: Other; Mean Difference (Final Values) = 16.3, 95% CI 2-sided [9.5 to 24.1]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); Vaccine Group Difference (aQIV - QIV) for B/Yamagata at Day 181; Test type: Other; Mean Difference (Final Values) = 46.4, 95% CI 2-sided [35.9 to 55.8]

13. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean HI Titers (GMTs) for Heterologous Influenza Strains (Day 1, Day 22, Day 181)
Description: Adjusted GMT, GMR and 95% CI were analyzed using ANCOVA with study specific covariates. Strains tested: A/H3N2 is Influenza A H3N2 Hong Kong/2014 Ab; B/Yamagata is Influenza B Phuket/2013 Ab
Time Frame: Day 1, Day 22, Day 181
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 155 | 138
titer
  Day 1: A/H3N2, Heterologous | 126.35 [83.7 to 190.8] | 48.02 [31.7 to 72.8]
  Day 22: A/H3N2, Heterologous: number analyzed (Participants) | 155 | 137
  Day 22: A/H3N2, Heterologous | 630.62 [515.0 to 772.2] | 402.54 [328.0 to 494.1]
  Day 181: A/H3N2, Heterologous | 304.10 [229.9 to 402.3] | 179.12 [134.9 to 237.7]
  Day 1: B/Yamagata, Heterologous | 30.29 [22.8 to 40.2] | 15.25 [11.5 to 20.3]
  Day 22: B/Yamagata, Heterologous: number analyzed (Participants) | 154 | 137
  Day 22: B/Yamagata, Heterologous | 196.27 [156.0 to 246.9] | 88.92 [70.6 to 112.0]
  Day 181: B/Yamagata, Heterologous: number analyzed (Participants) | 155 | 136
  Day 181: B/Yamagata, Heterologous | 69.60 [55.7 to 87.0] | 27.27 [21.8 to 34.1]
Statistical Analysis 1: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 1; Test type: Other; GMT Ratio = 2.63, 95% CI 2-sided [1.8 to 3.8]
Statistical Analysis 2: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 22; Test type: Other; GMT Ratio = 1.57, 95% CI 2-sided [1.3 to 2.9]
Statistical Analysis 3: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 181; Test type: Other; GMT Ratio = 1.70, 95% CI 2-sided [1.3 to 2.2]
Statistical Analysis 4: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for B/Yamagata at Day 1; Test type: Other; GMT Ratio = 1.99, 95% CI 2-sided [1.5 to 2.6]
Statistical Analysis 5: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 22; Test type: Other; GMT Ratio = 2.21, 95% CI 2-sided [1.8 to 2.7]
Statistical Analysis 6: Comparison: Adjuvanted Quadrivalent Influenza Vaccine (aQIV) vs Comparator Quadrivalent Influenza Vaccine (QIV); GMTr values between aQIV vs. QIV (ie, GMT[aQIV]:GMT[QIV]) for A/H3N2 at Day 181; Test type: Other; GMT Ratio = 2.55, 95% CI 2-sided [2.1 to 3.2]

14. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratios (GMR) for Heterologous Influenza Strains
Description: The GMR is the geometric mean of the fold increase in HI titer from Day 1 to Day 22 or Day 181. Adjusted GMT, GMR and 95% CI were analyzed using ANCOVA with study specific covariates. Strains tested: A/H3N2 is Influenza A H3N2 Hong Kong/2014 Ab; B/Yamagata is Influenza B Phuket/2013 Ab
Time Frame: Day 1, Day 22, and Day 181
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Adjuvanted Quadrivalent Influenza Vaccine (aQIV) | Comparator Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 155 | 138
ratio
  Day 22/Day 1: A/H3N2, Heterologous: number analyzed (Participants) | 154 | 137
  Day 22/Day 1: A/H3N2, Heterologous | 7.80 [6.4 to 9.6] | 4.98 [4.1 to 6.1]
  Day 181/Day 1: A/H3N2, Heterologous | 3.72 [2.8 to 4.9] | 2.19 [1.7 to 2.9]
  Day 22/Day 1: B/Yamagata, Heterologous: number analyzed (Participants) | 154 | 137
  Day 22/Day 1: B/Yamagata, Heterologous | 9.29 [7.4 to 11.7] | 4.21 [3.3 to 5.3]
  Day 181/Day 1: B/Yamagata, Heterologous: number analyzed (Participants) | 155 | 136
  Day 181/Day 1: B/Yamagata, Heterologous | 3.31 [2.7 to 4.1] | 1.30 [1.0 to 1.6]

ADVERSE EVENTS:
Time Frame: Serious AEs: SAEs were captured from day 1 through day 366. Non Serious AEs: Solicited local and systemic AEs were reported from day 1 through day 7 after vaccination. All unsolicited AEs were captured through day 366.
Description: All-cause mortality and non-serious AEs are reported for the Overall Safety Set (all subjects in the Solicited Safety Set and/or in the Unsolicited Safety Set). SAEs are reported for the Unsolicited Safety Set.
  Note: A total of 318 subjects were assigned to the aQIV arm; however, 1 subject in the aQIV arm incorrectly received QIV instead of aQIV and is included in the Comparator QIV arm for the safety analyses.
Arm/Group | aQIV | Comparator QIV
All-Cause Mortality (participants affected / at risk) | 0/317 | 0/290
Serious Adverse Events (participants affected / at risk) | 7/317 | 4/288
Other Adverse Events (participants affected / at risk) | 253/317 | 210/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=317) | Comparator QIV (N=288)
Right ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=317) | Comparator QIV (N=290)
Somnolence (Nervous system disorders) | 74 | 53
Influenza like illness (General disorders) | 24 | 30
Injection site erythema (General disorders) | 88 | 58
Injection site haemorrhage (General disorders) | 30 | 25
Injection site induration (General disorders) | 58 | 32
Injection site pain (General disorders) | 147 | 82
Pyrexia (General disorders) | 55 | 37
Eating disorder (Psychiatric disorders) | 55 | 30
Irritability (Psychiatric disorders) | 83 | 49
Diarrhoea (Gastrointestinal disorders) | 33 | 20
Vomiting (Gastrointestinal disorders) | 19 | 11
Otitis media (Infections and infestations) | 37 | 34
Pharyngitis streptococcal (Infections and infestations) | 16 | 6
Upper respiratory tract infection (Infections and infestations) | 32 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less